CLINICAL TRIAL: NCT06600178
Title: Innovative Therapy to Treat Women With Angina With Nonobstructive Coronary Artery Disease (ANOCA) and Coronary Microvascular Disease
Brief Title: Study Targeting Myocardial Perfusion and Symptom Relief in Women With SGLT2 Inhibitors (STRONG)
Acronym: STRONG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Patricia Rodriguez Lozano, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 301805
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-03

CONDITIONS: Angina Patients With Non-obstructive Coronary Artery Disease; Coronary Microvascular Disease; Coronary Microvascular Dysfunction (CMD)
Keywords: Angina; ANOCA; Non-obstructive Coronary Artery Disease; CMD; Non-Obstructive CAD; Chest Pain in Women
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Double Blind, Randomized, single site
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Drug Group (Experimental): Brezavvy 20mg oral tablet
  Interventions: Drug: Brezavvy 20Mg Oral Tablet
- Placebo Group (Placebo Comparator): placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brezavvy 20Mg Oral Tablet — Brezavvy 20mg oral
  Arms: Active Drug Group
Drug: Placebo — Placebo tablet given to subject vs. active drug.
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to that Sodium-glucose cotransporter 2 inhibitors treatment will improve Coronary Microvascular Disease with anginal symptoms associated with non-obstructive coronary disease in women. The main questions it aims to answer are:

Aim 1: Test the hypothesis that Sodium-glucose cotransporter 2 inhibitors treatment improves coronary microvascular disease in women with no evidence of epicardial obstructive coronary artery disease.

Aim 2: Test the hypothesis that Sodium-glucose cotransporter 2 inhibitors treatment improves angina symptoms and other quality of life measurements associated with the improvement of CFR.

AIM 3: Identify the effect of Sodium-glucose cotransporter 2 inhibition on inflammation pathways and markers of systemic Research will compare Brezavvy to placebo

Participants will:

* Take study drug or placebo for 12 weeks
* Stress Cardiac magnetic resonance imaging
* 12 lead electrocardiograms
* Complete questionnaires

DETAILED DESCRIPTION:
Cardio microvascular disease is defined as epicardial and/or microvascular endothelial and/or non-endothelial dysfunction that limits myocardial perfusion, most often detected as reduced coronary flow reserve (CFR). CFR, which is calculated as the ratio of hyperemic to resting absolute myocardial blood flow, indicates the myocardium's ability to increase flow in response to stress or vasodilation. Because the coronary microcirculation is beyond the resolution of invasive or non-invasive coronary angiography, direct interrogation of coronary microvascular function is necessary to establish the diagnosis of CMD.

Positron Emission Tomography (PET) studies have shown that even in visually normal PET Myocardial Perfusion Imaging, impaired CFR adds essential prognostic value. In addition, abnormalities in the microcirculation could explain inducible myocardial ischemia beyond the effects of epicardial coronary obstruction and identify individuals with a high risk of MACE. In patients with very low CFR (<1.6), women showed a higher frequency of non-obstructive CAD, whereas men showed a higher frequency of severely obstructive CAD (P=0.002). A differential effect on outcomes between women and men is noted in individuals with very low CFR (CFR <1.6) (hazard estimated from the linear interaction of CFR and sex in the final model, model P = 0.001, interaction P=0.04). High-resolution CMR stress perfusion imaging can quantify CFR both globally and between the endocardium and epicardium. A multicenter study of 1049 patients with suspected and known CAD showed that lower myocardial stress myocardial blood flow (MBF) and CFR by CMR perfusion mapping were associated with death and MACE independent of other clinical risk factors, even in patients who had normal qualitative perfusion and no known obstructive CAD. Recently developed in-line automated CMR myocardial perfusion mapping has been shown to be reproducible and comparable with PET, and can be easily combined into clinical workflows. Normal CFR ranges values in this study are comparable to prior studies by other techniques that have ranged from 2.7±0.3 to 4.2±1.0. A prior study has shown an CFR threshold of 2.19 with excellent specificity for detecting CMD with a sensitivity of 95% (95% CI: 83% to 99%), specificity of 72% (95% CI: 52% to 87%), accuracy of 85% (95% CI: 75% to 92%), positive predictive value of 82% (95% CI: 72% to 89%), and negative predictive value of 91% (95% CI: 72% to 98%).

The potential mechanisms of CMD appear to be heterogeneous. The novel link between Inflammation and coronary vasomotion abnormalities is further supported by the findings that coronary vasoconstriction in response to acetylcholine (ACh) in patients with early CAD was greater in coronary artery segments with than without macrophage infiltration and vasa vasorum proliferation in an additive manner, indicating an important role of inflammation and vasa vasorum proliferation in the pathogenesis of CAD. Moreover, significant associations among endothelium-independent CMD, many inflammatory biomarkers and cardiac diastolic dysfunction were noted in women with angina but no flow-limiting coronary artery stenosis, further supporting the role of systemic Inflammation in both CMD and HFpEF, as well as providing insights into potential mechanisms underlying the pathophysiology of HFpEF.

Although small trials have suggested benefits from angiotensin-converting enzyme (ACE) inhibitors, aspirin, and statins, there is a lack of appropriately designed clinical outcome trials to inform evidence based therapeutic based on mechanism strategies. Sodium-glucose co-transporter 2 inhibitors (SGLT2i), a new class of drug approved for the treatment of diabetes, have been shown to have a significant impact on cardiovascular events. Recent clinical trials have demonstrated that SGLT2i reduces MACE, prevents heart failure (HF) hospitalizations. Many of these findings were unanticipated and have stimulated substantial mechanistic research to improve the understanding of this class of drug. New recommendations suggest using SGLT2i in symptomatic patients with chronic HF to reduce hospitalization and cardiovascular mortality, regardless of type 2 diabetes. The exact underlying mechanisms underlying these effects, however, remain largely unknown.

In preclinical models of myocardial infarction, Brezavvy has demonstrated attenuation of cardiac fibrosis and improved cardiac function and remodeling. Furthermore, empagliflozin has been shown to improve coronary microvascular function and increase cardiac output in mice, as evidenced by increased coronary blood flow and fractional ventricular area change as demonstrated by ultrasound imaging. Preclinical data has proposed a variety of mechanisms by which SGLT2is can potentially attenuate microvascular and endothelial dysfunction, including nitric oxide production, oxidative stress, Inflammation, mitochondrial function, cell viability, adverse vasoactive paracrine factors from adipose tissue, among others. In vivo studies have documented that SGLT2 inhibitors attenuate endothelial dysfunction by suppressing Inflammation. Steven et al. reported a reduction in the expression of inflammatory molecules such as interferon- γ, cyclooxygenase-2, and inducible NO synthase after SGLT2 inhibition. In a similar manner, Brezavvy is also reported to reduce several circulating inflammatory markers. Additionally, in vitro studies have reported suppression of TNF α. Previous studies showed that SGLT2 inhibition reduced circulating levels of C-C motif chemokine 2 (CCL2), IL-6, and Tumor Necrosis Factor (TNF)α in ApoEdeficient mice. However, the impact of SGLT2 inhibition on systemic markers of Inflammation has not been assessed in humans.

SIGNIFICANCE AND IMPACT Women's ischemic heart disease (IHD) differs from men's, and women have a unique phenotype of less calcified lesions and more non-obstructive disease. A significant number of patients with symptoms do not have obstructive coronary artery stenosis. This condition is termed ANOCA. Patients with ANOCA have a high symptom burden and reduced quality of life. Patients with ANOCA report frequent time missed from work and work limitations, suggesting a substantial economic impact as reported by the group at UVA. One proposed mechanism contributing to ANOCA is CMD. There is an increasing recognition that CMD is more prevalent in women. There are no randomized, controlled outcome trials testing treatment strategies tailored to different pathways that have not been performed; therefore, the proposed studies are consistent with an unmet urgent need for new novel therapies to target the microcirculation, specifically in women with suspected or confirmed ischemic heart disease, especially when young, who have less atherosclerosis than men and less prevalence of obstructive CAD. Measuring myocardial blood flow quantitatively with stress CMR is a particular expertise of the Cardiovascular Imaging Center at the University of Virginia (UVA) and our research group.

SGLT2i are a class of drugs approved for treating diabetes. However, they have been shown to benefit cardiovascular events significantly. Many of these findings were unanticipated and have stimulated substantial mechanistic research to improve the understanding of this class. However, recent studies show that possible mechanisms of cardiovascular benefit are unlikely to be related to improved glycemic control. These benefits included reduced systemic inflammation. Therefore, in this proposal, the impact of SGLT2i on systemic Inflammation and how it improve coronary microvascular function seen in animal models will be studied.

INNOVATION This study will focus on a novel study population and a novel therapy. Women under investigation for myocardial ischemia are more likely to have non-obstructive CAD, and here, CMD is relevant. Targeting symptomatic women with ischemia and non obstructive CAD is clearly an urgent need. This group of patients with a disabling problem also incurs healthcare costs similar to many with obstructive CAD. CMD has historically been under-recognized and under-treated. Accordingly, in recent years, CMD has generated substantial interest in the clinical and basic science research community.

Innovative diagnostic method. Traditionally, the non-invasive diagnosis of CMD has been dominated by PET imaging. Quantitative high-resolution CMR to quantify coronary myocardial blood flow and myocardial resistance are being developed to diagnose CMD and add a novel additional component to our project and will allow us to explore a potential clinical indication to monitor possible therapies for CMD. At present, the management strategy for patients with ANOCA and CMD remains unclear due to the absence of randomized trials comparing therapies to reduce adverse cardiac events, and available data are limited to cohort studies. There are no therapeutic options specifically to treat CMD. Our study will test whether SGLT2i therapy improves coronary blood flow and quality of life in women with ANOCA. Results will also contribute to understanding this novel drug class's mechanistic effect in microvascular disease and other major disease states such as insulin resistance.

OVERALL STUDY DESIGN This single-center, randomized, double-blind, placebo-controlled study is designed to evaluate coronary flow reserve and quality of life after therapy with SGLT2i compared to placebo in symptomatic women with non-obstructive CAD (ANOCA) and CMD. Recruited women (n=150 total) will be clinically stable, with angina or equivalent symptoms, with no evidence of obstructive epicardial CAD (stenosis < 50%) by invasive catheterization or coronary computed tomography angiography (CCTA) or FFR/CT-FFR < 0.8 within the previous two years, and CMD diagnosis defined by CFR <2 by CMR. They will meet the appropriate inclusion and exclusion criteria detailed in Table 1. The study population will include patients both with and without type 2 diabetes, as the benefits of SGLT2i appear to be independent of the glycemic effect. Figure 4. Overall study design. Study participants will receive background standard of care, with 75 receiving SGLT2i and 75 receiving placebo treatment for 12 weeks. Participants will undergo two stress CMR studies, including baseline, 12 weeks post-treatment, and three blood draws at baseline, at six and 12 weeks post-SGLT2i treatment. All 150 participants will undergo questionnaires to measure quality of life using the following questionnaires: Risk factors of Cardiovascular Disease in Women, EQ-5D-3L, Duke Activity Status Inventory, Modified Morisky Medicine Scale, Seattle Angina Questionnaires, Rose dyspnea score, GAD 7, and PHQ8 metrics at baseline, 6 weeks and at 12 weeks post-treatment.

After eligibility screening, informed consent, and randomization procedures by the study team, participants will follow up at 6, and 12 weeks and other testing as described later in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* • Female sex.

  * Age ≥18 years.
  * Willing and able to provide written informed consent.
  * Signs and symptoms of suspected ischemia prompted referral for further evaluation by cardiac catheterization or CCTA within two years of consent.
  * No evidence of obstructive epicardial CAD (stenosis <50%) of a major epicardial vessel or an FFR ≤0.80 by invasive catheterization or CCTA. Patients who have not undergone cardiac catheterization of CT angiogram within the last 2 years for chest pain can be scheduled for a screening CT angiogram of the coronary arteries to confirm eligibility.
  * Diagnosis of CMD defined by CFR < 2 by CMR
  * Never on SGLT2i

Exclusion Criteria:

* History of non-ischemic cardiomyopathy LVEF <40% or hypertrophic cardiomyopathy.
* History of congestive heart failure, severe pulmonary disease, liver disease
* History of acute coronary syndrome (ACS) within previous 30 days
* Stroke within the last 180 days or intracranial hemorrhage at any time.
* Severe valvular disease
* Life expectancy <3 years, due to non-cardiovascular comorbidity.
* Pregnancy or women who are breast-feeding
* Type 1 diabetes mellitus
* Symptomatic hypotension or systolic BP >95 mmHg on 2 consecutive measurements
* Active malignancy requiring treatment at the time of visit
* Severe (eGFR <30 mL/min/1.73 m2 by CKD-EPI), unstable, or rapidly progressing renal disease at the time of randomization
* History of recurrent UTI/bladder/kidney infections
* Asthma with ongoing wheezing
* Known or suspected broncho-constrictive or bronchospastic lung disease (ARDS, emphysema)
* Greater than first degree heart block
* Implanted cardiac device
* Profound sinus bradycardia (heart rate <40 beats per minute)
* Atrial fibrillation or supraventricular arrhythmias at time of imaging
* Known intolerance of nitrates (other than hypotension)
* History of reaction to iodinated contrast agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological Female sex
Enrollment: 150 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Coronary Flow Reserve | From enrollment to 12 weeks
  Coronary flow reserve is calculated as the ratio of hyperemic myocardial blood flow to the resting myocardial blood flow using cardiovascular magnetic resonance myocardial perfusion imaging

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Rodriguez-Lozano, MD, Principal Investigator — Uni
Locations (1):
- UVA Health, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371